CLINICAL TRIAL: NCT01996995
Title: Laser Therapy for Onychomycosis in Patients Wih Diabetes at Risk for Diabetic Foot Complications
Acronym: LASER-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Henk Bilo, MD, MD PhD, Medical Research Foundation, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL46084.075.13; NL46084.075.13 (Other Grant/Funding Number: NL46084.075.13)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nd:YAG laser pulse therapy (Experimental): Nd:YAG laser pulse therapy Patients are treated with laser session in week 0, 2, 4, and 12. The settings are; 1064 nm, spot size 3 mm, 20 J /cm2, 5 Hz, power 10 W, pulse duration 132 millisecond. A maximum of two sequential sessions (one session on the horizontal and one the vertical passing) will be applied to eliminate potential safety issues in those patients with a lack protective sensibility.
  Interventions: Device: Nd:YAG laser pulse therapy
- Sham (Sham Comparator): Sham treatment Patients are treated with a sham session in week 0, 2, 4, and 12. The study settings are similar to the laser except the laser beam. Because the patient is also blinded, they can't see the procedure. The sound and the beeps are audible similar to the laser treatment.
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: Nd:YAG laser pulse therapy
  Other Names: S30 PODYLAS
  Arms: Nd:YAG laser pulse therapy
Device: Sham procedure — Sham procedure
  Arms: Sham

SUMMARY:
In a sham controlled double-blind trial we aim to establish the efficacy and safety of local application of laser therapy in patients with diabetes with onychomycosis and risk factors for diabetes related foot complications. Onychomycosis leads to thickened and distorted nails, which in turn leads to increased local pressure. The combination of onychomycosis and neuropathy or peripheral arterial disease (PAD) increases the risk of developing diabetes related foot complications. Usual care for high-risk patients with diabetes and onychomycosis is completely symptomatic with frequent skiving and clipping of the nails. No effective curative local therapies exist and systemic agents are often withheld due to concerns for side effects and interactions.

Aim: The primary aim is to evaluate the efficacy of 4 sessions N-YAG 1064nM laser application on the one-year clinical and microbiological cure rate in a randomised, double-blinded sham-controlled design with blinded outcome assessment.

Study population: Patients with diabetes mellitus, with an increased risk for diabetic foot ulcers.

Intervention: local laser treatment from a podiatrist and the other group receives treatment according to a control procedure. The laser procedure will be performed as a sham procedure by a second podiatrist.

Main study parameters/endpoints: The effect of 4 sessions of laser therapy on cure rate (clinical and microbiological) after one year.

DETAILED DESCRIPTION:
Setting of the study: Hospital, outpatient departments (Foot clinic, Isala, Zwolle)

Inclusion criteria: Patients with clinical suspicion and microbiologic confirmation of onychomycosis , diagnosis of T1DM or T2DM, 18 years or older, at risk for diabetic foot ulcers defined by a modified Simm's classification score 1 or 2 with either neuropathy or PAD, nail involvement of at least 25% of the target nail.

Exclusion criteria: no microbiologic confirmation, Simms' classification score 3, the presence or history of diabetic foot ulcers, ischemic pain, ankle brachial index < 0.9, patients receiving dialysis, severe renal insufficiently (eGFR below 30 ml/min), a documented toe pressure below 50 mmHg, use of systemic or topical antifungal agents 3 months prior to inclusion, use of immunosuppressive drugs, presence of psoriasis, lichen planus, or other abnormalities that could result in clinically abnormal toenails, a history of epilepsy and insufficient knowledge of the Dutch language. Patients with a dark skin color (Fitzpatrick 4 and 5) are excluded since dark skin color is associated with dark nails, which theoretically leads to increased temperatures during laser application

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Over 18 years old
* Clinically suspicion with microbiologic confirmation of onychomycosis
* Patient is at risk for diabetic foot ulcers defines as Simms score 1, 2 .

Exclusion Criteria:

* Patients without the microbiological confirmation of fungal nail infection
* Patients with an active or history of a diabetic foot ulcer
* Patients who used systemic or topical anti fungal agents during the preceding 3 months
* Patients with ischemic rest pain
* Patients with ankle brachial index < 0.9
* Patients with a documented toe pressure below 50 mmHg
* Patients receiving dialysis, severe renal insufficiently (eGFR below 30 ml/min)
* Patients with an insufficient knowledge of the Dutch language to understand requirements of the study
* Patients with a dark skin color (Fitspatrick 4 and 5)
* Patients who uses immunosuppressive medication
* Patient suffering from nail psoriasis , lichen planus, or other abnormalities that could result in clinically abnormal toenails.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
complete cure of the target nail | outcome measured after 1 year
  after one year the clinical and microbiological cure rate of the target nail will be compared with usual care in the placebo group.

SECONDARY OUTCOMES:
Microbiological cure of the target nail | outcome measured after 1 year
  Patient with a negative microbiologic results of the target nail at week 52 will be regarded as having a microbiological cure. Patients with negative microbiological results at week 30 and positive microbiologic results at week 52 will be regarded as having a second infection. Patients with positive microbiologic results (with the same species) at week 30 and positive results at week 52 (the same species) will be regarded as treatment failure.
Complete clinical cure of the target nail | outcome measured after 1 year
  Complete cure is defined as a completely normal nail, or negative microbiological results in case minor abnormalities are present.
Markedly clinically improved target nail | outcome measured after 1 year
  A markedly improved nail is defined as a nail with less than 10% abnormalities without hyperkeratosis after 52 weeks in nails that were affected more than 10% of the surface area.
Onychomycosis severity index below 6 (in patients with scores >6 at study entry) of the target nail | outcome measured after 1 year
Complete clinical cure of all affected toes | outcome measured after 1 year
Change in quality of life | outcome measured after 1 year
  WHO-5 and NailQol questionnaires are taken at baseline and week 52. Translated disease specific questionnaire; NailQol
Change surface healthy target nail / all clinically infected toes patients free of hyperkeratosis | outcome after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: H.J.G. Bilo, professor MD, Study Director — Isala Diabetes Centre, Zwolle; Nanne Kleefstra, MD PhD, Study Director — Isala Diabetes Centre,Zwolle; G.W.D. Landman, MD PhD, Principal Investigator — Isala Diabetes Centre, Zwolle; Leonie Nijenhuis - Rosien, Bsc, Principal Investigator — Isala Diabetes Centre, Zwolle
Locations (1):
- Isala Diabetes Centre, Isala Hospital, Zwolle, Netherlands

REFERENCES:
- [Derived] Nijenhuis-Rosien L, Kleefstra N, Wolfhagen MJ, Groenier KH, Bilo HJ, Landman GW. Laser therapy for onychomycosis in patients with diabetes at risk for foot complications: study protocol for a randomized, double-blind, controlled trial (LASER-1). Trials. 2015 Mar 22;16:108. doi: 10.1186/s13063-015-0622-4. PMID 25872590
- Available data/document: Study Protocol — http://trialsjournal.biomedcentral.com/articles/10.1186/s13063-015-0622-4